CLINICAL TRIAL: NCT02519543
Title: Treating Insulin Resistance to Improve Outcome in Refractory Bipolar Disorder: a Randomized, Double-blind, Placebo-control Study of the Efficacy of Metformin in Patients With Insulin Resistance and Non-remitting Bipolar Illness
Brief Title: Treating Insulin Resistance as a Strategy to Improve Outcome in Refractory Bipolar Disorder
Acronym: TRIO-BD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cynthia Calkin (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Cynthia Calkin, Cynthia Calkin, Associate Professor, Dalhousie University, Nova Scotia Health Authority, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRIO-BD-100
Record Dates: First submitted 2015-08-03; First posted 2015-08-11 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Bipolar Disorder
Keywords: insulin resistance
MeSH Terms: conditions — Bipolar Disorder; Insulin Resistance | interventions — Sugars; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo comparator to be given twice daily, once with breakfast and once with supper
  Interventions: Drug: Placebo
- Metformin (Experimental): Metformin 2000 mg daily to be given as follows: 1000 mg with breakfast and 1000 mg with supper
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo — Placebo to be given twice daily, once with breakfast and once with supper
  Other Names: sugar pill
  Arms: Placebo
Drug: Metformin — Active experimental drug to be given twice a day, 1000 mg with breakfast and 1000 mg with supper
  Other Names: Metformin Hydrochloride
  Arms: Metformin

SUMMARY:
In a previous study by Dr. Calkin, the principal investigator of this study, persons with bipolar disorder and either type II diabetes or insulin resistance were found to experience more severe symptoms of bipolar illness and a lower response to treatment, compared to persons with bipolar disorder who did not have type II diabetes or insulin resistance. To further explore these findings, the investigators have developed this study to see if treating insulin resistance (using metformin, a drug used to improve the body's use of insulin) may also help improve the symptoms of bipolar illness.

DETAILED DESCRIPTION:
This is a 26-week randomized, double-blind, parallel group prospective study of the effectiveness of treating insulin resistance (IR) to improve mood in patients with IR and treatment-resistant bipolar depression (TRBD). The investigators will compare the effects of treating IR (with metformin) versus placebo on outcome in each patient. The primary outcome will be change in Montgomery-Ǻsberg Depression Rating Scale (MADRS) scores. Patients' current optimized mood stabilizing treatment as usual (TAU, according to the Canadian Network for Mood and Anxiety Treatments [CANMAT] or American Psychiatric Association [APA] guidelines) must remain unchanged for a period of at least 4 weeks prior to and throughout the study. Patients will undergo a baseline assessment and then be randomized to treatment with metformin or placebo with titration to full dose after 2 weeks. Patients will remain on full treatment for 24 weeks thereafter (total trial duration of 26 weeks for each patient). In those patients with TRBD assigned to treatment with the insulin sensitizer metformin, a significant improvement in depression symptoms will be mediated by the conversion of IR to insulin sensitivity.

Subjects: We aim to enrol 110 subjects with IR and TRBD from 2 sites: the primary site in Halifax, Nova Scotia, Canada, and a second site in Pittsburgh, Pennsylvania, USA.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. diagnosis of BD I or II
3. non-remitting BD as defined by the presence of mood symptoms of at least moderate severity, indicated by a MADRS score ≥ 15 despite being on optimal treatment according to the CANMAT/APA guidelines
4. HOMA-IR ≥ 1.8, indicating IR (subjects will have FPG and FSI testing done to determine whether they have IR or T2D)
5. current episode of depression 4 weeks or longer in duration
6. on a stable optimal dose of mood stabilizing treatment for at least 4 weeks prior to study entry

Exclusion Criteria:

1. Diagnoses of organic mood disorder, mood disorder not otherwise specified, alcohol dependence, T1D or T2D
2. presence of rapid cycling (by DSM-5 criteria), mania, (indicated by a Young Mania Rating Scale [YMRS] score > 15), or suicide ideation (current score of 5 on the Suicidal Ideation section of the Columbia-Suicide Severity Rating scale [C-SSRS])
3. patient receiving metformin < 2 weeks prior to study entry
4. metformin allergy or sensitivity
5. metformin contraindicated where liver function tests > three times the upper limit of normal, estimated glomerular filtration rate (eGFR) < 30, CBC revealing megaloblastic anemia or pre-existing untreated B12 deficiency
6. pregnancy or breastfeeding
7. lactose intolerance, diagnosed by a physician
8. chronic use of narcotic medications
9. patient lacks full capacity to consent to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Montgomery-Ǻsberg Depression Rating Scale (MADRS) | 14 weeks
  Using this scale, we will study the effect of treating insulin resistance (IR) on bipolar depression symptoms after 14 weeks of study drug treatment. We will assess whether the effect of metformin on improvement in MADRS scores at week 14 is mediated by conversion of IR to insulin sensitivity (determined using Homeostatic Model Assessment - Insulin Resistance, i.e. HOMA-IR).

SECONDARY OUTCOMES:
Montgomery-Ǻsberg Depression Rating Scale (MADRS) | 26 weeks
  Using this scale, we will assess whether the effect of treating IR on bipolar depression symptoms is sustained up to 26 weeks.
Montgomery-Ǻsberg Depression Rating Scale (MADRS) | 14 and 26 weeks
  Using this scale, we will assess whether treating IR results in a ≥ 30% improvement in bipolar depression symptoms after 14 weeks and 26 weeks of study drug treatment.
Inventory of Depressive Symptomatology-Self Rating (IDS-SR) | 14 and 26 weeks
  We will examine the effect of treating IR on mood and anxiety symptoms using this rating scale.
Young Mania Rating Scale (YMRS) | 14 and 26 weeks
  We will examine the effect of treating IR on mania symptoms using this rating scale.
Hamilton Anxiety Rating Scale (HAM-A) | 14 and 26 weeks
  We will examine the effect of treating IR on mood and anxiety symptoms using this rating scale.
Clinical Global Impression modified for use in Bipolar Disorder (CGI-BP) | 14 and 26 weeks
  We will use this scale to assess the effect of treating IR on overall psychiatric morbidity and severity of illness.
Global Assessment of Functioning (GAF) | 14 and 26 weeks
  We will use this scale to assess the effect of treating IR on overall psychiatric morbidity and severity of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Calkin, MD FRCPC, Principal Investigator — Nova Scotia Health Authority; Roy Chengappa, MD FRCPC, Principal Investigator — Western Psychiatric Institute and Clinic, University of Pittsburgh Medical Center
Locations (2):
- Western Psychiatric Institute and Clinic, University of Pittsburgh Medical Center, University of Pittsburgh, Pittsburgh, Pennsylvania, United States
- Nova Scotia Health Authority - Dept. of Psychiatry, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calkin CV, Ruzickova M, Uher R, Hajek T, Slaney CM, Garnham JS, O'Donovan MC, Alda M. Insulin resistance and outcome in bipolar disorder. Br J Psychiatry. 2015 Jan;206(1):52-7. doi: 10.1192/bjp.bp.114.152850. Epub 2014 Oct 16. PMID 25323142
- [Background] Ruzickova M, Slaney C, Garnham J, Alda M. Clinical features of bipolar disorder with and without comorbid diabetes mellitus. Can J Psychiatry. 2003 Aug;48(7):458-61. doi: 10.1177/070674370304800705. PMID 12971015
- [Background] Calkin CV, Gardner DM, Ransom T, Alda M. The relationship between bipolar disorder and type 2 diabetes: more than just co-morbid disorders. Ann Med. 2013 Mar;45(2):171-81. doi: 10.3109/07853890.2012.687835. Epub 2012 May 24. PMID 22621171
- [Derived] Calkin CV, Chengappa KNR, Cairns K, Cookey J, Gannon J, Alda M, O'Donovan C, Reardon C, Sanches M, Ruzickova M. Treating Insulin Resistance With Metformin as a Strategy to Improve Clinical Outcomes in Treatment-Resistant Bipolar Depression (the TRIO-BD Study): A Randomized, Quadruple-Masked, Placebo-Controlled Clinical Trial. J Clin Psychiatry. 2022 Feb 1;83(2):21m14022. doi: 10.4088/JCP.21m14022. PMID 35120288
- See also: The risk of insulin resistance and type 2 diabetes mellitus in bipolar disorder — https://apps.webofknowledge.com/full_record.do?product=UA&search_mode=GeneralSearch&qid=1&SID=2CRUvkzBT6AQyUenrvK&page=2&doc=11
- See also: Are comorbid insulin resistance and type II diabetes risk factors for refractory bipolar illness? — http://ac.els-cdn.com.ezproxy.library.dal.ca/S0924977X13705789/1-s2.0-S0924977X13705789-main.pdf?_tid=234a7e9a-3c2e-11e5-ace4-00000aab0f01&acdnat=1438860636_5aecad769a45feae96b677c0ccb908cc